CLINICAL TRIAL: NCT04834960
Title: Missed Opportunities for Vaccine Equity
Acronym: MOVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Post Graduate Institute of Medical Education and Research, Chandigarh (Other); Aminu Kano Teaching Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: I1429
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Under-vaccinated
Keywords: vaccination; under-vaccination; missed opportunities for vaccination
MeSH Terms: interventions — Vaccination

STUDY DESIGN:
Intervention Model Description: This is a 'pre-post' study design, where the intervention is designed and implemented by the regular non-research clinical staff. This intervention has four components that are described in the 'intervention' section.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MOV Intervention (Other): Pre-intervention and post-intervention design
  Interventions: Other: Minimizing Missed Opportunities for Vaccination (MOV)

INTERVENTIONS:
Other: Minimizing Missed Opportunities for Vaccination (MOV) — This bundle of interventions has four components that include: (1) Disseminate (vaccination awareness among healthcare providers and child caregivers); (2) Document (vaccination status); (3) Deploy (vaccines); and (4) Discharge (provide advice/referrals for catch-up and routine vaccinations).

SUMMARY:
Despite the overwhelming impact of vaccines on child health and the tremendous progress in vaccine coverage globally, challenges of vaccine inequities persist. Missed opportunities for vaccination (MOV) is defined as any contact with health services by an individual who is eligible for vaccination which does not result in the recommended vaccines being given. This is common in several countries, and it presents a window of opportunity to provide vaccine services to those vulnerable children accessing healthcare facilities.

The overall purpose of this project is to reduce missed opportunities for vaccinations by targeting hospitalized children who are vulnerable to poor health outcomes, but who are also within easy access of the healthcare system. The research team proposes implementing the Missed Opportunities for Vaccination Equity (MOVE), an intervention to improve timeliness and coverage of vaccination, and increase demand for vaccination services, through a combination of sensitization of children's caregivers and health workers, manual vaccination data capture in the ward, and re-purposed vaccination resources. The strategy engages key stakeholders in the design of the intervention through a co-creation workshop; their involvement in the design and execution of the intervention will improve sustainability in the long-term. This intervention builds on existing healthcare systems, and, when scaled up, can target inequities in vaccination coverage in the general population, without placing additional strain on the healthcare system in terms of workforce or financial resources.

DETAILED DESCRIPTION:
This pilot project is structured as a pre-post analysis of an implementation strategy to address missed opportunities for vaccination (MOV) among hospitalized children in India and Nigeria. India and Nigeria have similar rates of missed opportunities for vaccinations, and similar discrepancies with monitoring vaccination records when a child is in the hospital. The research team intends to collect the same pre-data in both India and Nigeria, implement the same intervention in both countries, and collect the same post-data in both study sites.

The pre-intervention, intervention, and post-intervention, are all described below.

Pre-Intervention period: The first three months of the project constitute the pre-intervention period, and they will consist of a situational analysis which will assess the burden of MOV as well as the barriers and facilitators for reducing MOV. Eligible participants will be enrolled after providing informed consent. Procedures would include verifying vaccination cards and medical records at admission and at discharge, conducting in-depth interviews with parents or caregivers during the hospital course, and administering structured questionnaires to hospital healthcare personnel crucial to hospitalized child care and provision of vaccinations.

Intervention: This will begin with a co-creation workshop where the results of the pre-intervention period will be discussed, and the MOV intervention will be implemented. In summary, the intervention will include four components which are: (1) Disseminate (vaccination awareness among healthcare providers and child caregivers); (2) Document (vaccination status); (3) Deploy (vaccines); and (4) Discharge (provide advice/referrals for catch-up and routine vaccinations).

Using a human-centered design approach, the research team will design an intervention, endorsed by local healthcare providers and stakeholders, which will be implemented primarily by the existing hospital healthcare staff. Research staff will play a role in data collection for monitoring purposes, but will not play a role in implementing the intervention.

Post-Intervention period: Ongoing data collection after the MOV intervention is initiated and continued, will constitute the 'post-intervention' period. During this period, data collectors will collect the same data that is being collected in the pre-intervention. The research team intends to compare the results of our pre and post intervention data, to determine if this intervention has reduced the amount of children who are missed for vaccinations.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages 0-23 months who are admitted into the emergency or inpatient unit of the hospital
* Caregiver has access to the child's vaccination card or has direct knowledge of the child's vaccination history
* Caregiver willing to provide informed consent for the study

Exclusion Criteria:

* Health condition that precludes the use of vaccines such as a primary or secondary immune deficiency, such as HIV, malignancy requiring chemotherapy, or ongoing steroid therapy
* Allergies or contraindications to any vaccine (or component thereof) in the national schedule

Ages: 0 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 900 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-09-16 (Actual)

PRIMARY OUTCOMES:
Proportion of Children Fully Vaccinated Hospital Discharge | time of admission to discharge (about 1-2 weeks)
  The number fully vaccinated at admission + number given catch-up vaccination while in hospital, and up to the date at discharge / the number of all enrolled children. This outcome measures the desired outcome of full vaccination coverage among children who pass through in-patient health facilities. This is the main outcome of interest and will be compared in the pre-intervention and post-intervention phases.
Partially Vaccinated or Un-vaccinated Children at Admission | time of admission to discharge (about 1-2 weeks)
  This is the proportion of those children who are under-vaccinated at hospital admission.
Proportion of Under-Vaccinated children Deemed "Missed Opportunities of Vaccination" | time of admission to discharge (about 1-2 weeks)
  The number of eligible children who do not receive their due catch-up vaccines prior to hospital discharge / the number of children identified as under-vaccinated at hospital admission.
Proportion of all Enrolled Children at Admission Given Vaccination Advice | time of admission to discharge (about 1-2 weeks)
  The number of all enrolled children at admission who get vaccination-related advice and/or referrals during the hospital stay / the number of all enrolled children participating in the study.
Proportion of Incompletely Vaccinated Children Caught up After Discharge | time of admission (about 1-2 weeks) to 1 month post discharge
  The number of incompletely vaccinated children at hospital discharge who get caught up on vaccinations within 1-4 weeks of hospital discharge / the number of children identified as under-vaccinated at hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Shet, MD, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (2):
- Post Graduate Institute of Medical Education and Research, India (PGIMER), Chandigarh, India
- Aminu Kano Teaching Hospital, Kano, Kano State, Nigeria

IPD SHARING:
Plan to Share IPD: No